CLINICAL TRIAL: NCT03150368
Title: Safety of Extended Use of ModraDoc006/r in Patients With Advanced Solid Tumours
Brief Title: Extended Use of ModraDoc006/r
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Modra Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N17DEX
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Advanced Solid Tumours

STUDY DESIGN:
Intervention Model Description: After completion of a phase 1 trial with ModraDoc006/r, patients are able to continue weekly treatment with oral docetaxel (ModraDoc006) in combination with ritonavir, for as long as safe clinical benefit from the treatment is experienced, as judged by the treating oncologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ModraDoc006/r (Experimental): Weekly ModraDoc006/r treatment as ModraDoc006 (oral docetaxel) 10mg tablets combined with ritonavir 100mg tablets
  Interventions: Drug: ModraDoc006/r

INTERVENTIONS:
Drug: ModraDoc006/r — Treatment with weekly ModraDoc006 (oral docetaxel) 10mg tablets in combination with ritonavir 100mg tablets
  Other Names: oral docetaxel formulation

SUMMARY:
This is a study for extended use of ModraDoc006/r in patients with advanced solid tumours, available after completed treatment in one of the phase I trials with ModraDoc006/r. The primary goal is to explore the safety of extended use.

DETAILED DESCRIPTION:
This is an open label extended use programme, designed to make extended use treatment with weekly ModraDoc006/r available for patients who completed treatment in one of the phase I trials with ModraDoc006/r, who might have clinical benefit of continued treatment with the oral docetaxel formulation.

Patients will receive oral docetaxel (as ModraDoc006 10 mg tablets) and ritonavir (100 mg tablet) once- or bi-daily, once a week in a fasted condition. Treatment can be continued weekly as long as the patient experiences clinical benefit from the treatment as judged by the treating oncologist, unless unacceptable toxicity despite dose modifications and supportive measures occurs.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of cancer
2. Patients who might benefit from a weekly (oral) docetaxel regime as judged by the treating oncologist.
3. Patients who received treatment with ModraDoc006/r with acceptable safety (as judged by the PI; for criteria see below in section 3 of exclusion criteria) in phase I trials with ModraDoc006/r, including (but not limited to) the N15FED (food-interaction study), N16AED (absorption-excretion study), N16DOL (normal or impaired liver function). A maximum delay of 21 days between the last dose in the previous phase I trial and the first dose in the N17DEX is allowed.
4. Age ≥ 18 years
5. WHO performance status of 0, 1 or 2;
6. Minimal acceptable laboratory values defined as:

   1. ANC of ≥ 1.5 x 109 /L
   2. Platelet count of ≥ 100 x 109 /L
   3. Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula)
   4. Hepatic function as defined by serum bilirubin ≤ 2 x ULN, ALAT and ASAT ≤ 5.0 x ULN, except for patients who have been treated in the N16DOL study.
7. Negative pregnancy test (urine/serum) for female patients with childbearing potential, assessed at the screening visit of the previous phase I trial with ModraDoc006/r.
8. Able and willing to swallow oral medication

Exclusion Criteria:

1. Concomitant use of MDR and CYP3A modulating drugs such as Ca+-entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, quinine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications; other protease inhibitors, (non) nucleoside analogs, St. John's wort or macrolide antibiotics.
2. Symptomatic brain metastases or leptomeningeal metastases. Patients with brain metastases are allowed if they received adequate treatment, are asymptomatic in the absence of corticosteroid therapy and anticonvulsant therapy for at least 6 weeks. Radiotherapy for brain metastases must have been completed at least 4 weeks prior to start of study treatment.
3. Clinically significant safety issues during previous therapy with ModraDoc006/r as judged by the PI, which cannot be solved by dose reduction and/or treatment delay.
4. Unreliable contraceptive methods. Both men and women using ModraDoc006/r must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms).
5. Anti-cancer therapy or any treatment with investigational drugs other than ModraDoc006/r between the completion of the phase I trial with ModraDoc006/r and the start of extended use of ModraDoc006/r Palliative radiation on limited field is allowed.
6. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients. Patients with a known history of hepatitis B or C.
7. Bowel obstructions or motility disorders that may influence the resorption of drugs as judged by the treating physician.
8. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance; Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
The hematological and non-hematological toxicity profile of oral docetaxel in combination with ritonavir | Safety and tolerance will be evaluated during the complete study treatment until 28 days after the last intake, using the CTCAE v.4.03 grading system
  The number of CTCAE v.4.03 grade 3-4 toxicities during treatment with ModraDoc006/r

CONTACTS AND LOCATIONS:
Overall Officials: Serena Marchetti, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No